CLINICAL TRIAL: NCT05276713
Title: A Single-center Study of the Outcome of Tucidinostat-Based Therapy in Hormone Receptor-Positive Metastatic Breast Cancer Patients Previously Treated With CDK4/6 Inhibitor Therapy
Brief Title: Outcome of Tucidinostat-Based Therapy in HR+ Metastatic Breast Cancer Patients Previously Treated With CDK4/6 Inhibitor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Breast-Chi-2022
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tucidinostat-based therapy: 30 mg tucidinostat was given orally(as six 5 mg tablets per day) twice a week (either, Monday and Thursday, Tuesday and Friday, or Wednesday and Saturday) for 4 consecutive weeks in a 4-week cycle.The endocrine drugs combined with tucidinostat were given based on previous treatment.Patients received tucidinostat-based treatment until disease progression or intolerable adverse events.
  Interventions: Drug: Tucidinostat

INTERVENTIONS:
Drug: Tucidinostat — Tucidinostat in combination with endocrine drugs
  Other Names: Chidamide

SUMMARY:
To evaluate the efficacy of tucidinostat-based therapy in hormone receptor-positive metastatic breast cancer patients previously treated with CDK4/6 inhibitor therapy in the real world.

DETAILED DESCRIPTION:
Cyclin-dependent kinase (CDK) 4/6 inhibitors have changed the treatment pattern of patients with hormone receptor-positive HER2-negative advanced breast cancer significantly prolongling patients'PFS and OS,but there is no optimal therapy after its progression.Tucidinostat (formerly known as chidamide) is an oral subtype-selective histone deacetylase inhibitor, ACE trial demonstrated that tucidinostat plus exemestane improved PFS compared with placebo plus exemestane in HR+,MBC patients that progressed after previous endocrine therapy,only 7 patients enrolled in the trial had previously received CDK4/6 inhibitors.The aim of this trial is to evaluate the efficacy of tucidinostat-based therapy in hormone receptor-positive metastatic breast cancer patients previously treated with CDK4/6 inhibitor therapy in the real world.

ELIGIBILITY:
Inclusion Criteria:

* 1.woman, age > 18 years old 2.Diagnosed with HR+/HER2- Metastatic Breast Cancer 3.Patients received tucidinostat-based therapy after progression on CDK4/6 inhibitor 4.Complete medical history was available

Exclusion Criteria:

* 1.Medical history was incomplete

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to International Classification of Diseases-10, ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Tao wang, Study Director — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No